CLINICAL TRIAL: NCT06740032
Title: Comparison of the Acute Effects of Auricular Vagus Nerve Stimulation and Deep Breathing Exercise on the Autonomic Nervous System Activity and Biomechanical Properties of the Muscle in Healthy People
Brief Title: Comparison of the Acute Effects of Auricular Vagus Nerve Stimulation and Deep Breathing Exercise
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Gelisim University (Other)
Collaborators: Bahçeşehir University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: VNS06.01.2022/01
Record Dates: First submitted 2024-11-29; First posted 2024-12-18 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Vagus Nerve Stimulations
Keywords: Auricular vagus nerve stimulation; deep breathing exercises

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- autonomic function (Active Comparator)
  Interventions: Other: Transcutaneous vagus nerve stimulation; Other: Deep breath exercise
- somatic function (Active Comparator)
  Interventions: Other: Transcutaneous vagus nerve stimulation; Other: Deep breath exercise

INTERVENTIONS:
Other: Transcutaneous vagus nerve stimulation — Investigation of the effects of vagus nerve stimulation on the autonomic and somatic systems together
Other: Deep breath exercise — Investigation of the effects of vagus nerve stimulation on the autonomic and somatic systems together

SUMMARY:
The goal of this clinical trial is to investigate whether vagus stimulation and breathing exercises are more effective in healthy adults.

Are vagal stimulation and breathing exercises effective on autonomic functions and the somatic system in healthy adults? Participants' results for autonomic functions and somatic system will be compared for both groups.

ELIGIBILITY:
Inclusion Criteria:

* could read and write Turkish

Exclusion Criteria:

* being 18 years or older having no known acute or chronic disease, and no previous treatment with vagus nerve stimulation

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2022-02-27 (Actual); Primary Completion 2022-06-12 (Actual); Study Completion 2022-08-28 (Actual)

PRIMARY OUTCOMES:
HRV results | 5 minutes
  Measuring autonomic values for 5 minutes
Muscle Natural Oscillation Frequency | 5 minutes
  Biomechanical measurements of specific muscles
Muscle Dynamic Stiffness [N/m] | 5 minutes
  measured using the myoton device
Mechanical Stress Relaxation Time [ms] | 5 minutes
  measured using the myoton device

SECONDARY OUTCOMES:
Perceived stress scale | 5 minutes
  Evaluation of stress levels with the specified questionnaire
Pulse rate | 5 minutes
  Measuring with a sphygmomanometer
blood pressure | 5 minutes
  Measuring blood pressure with a sphygmomanometer

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Gelisim University, Istanbul, Avcılar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://tez.yok.gov.tr/UlusalTezMerkezi/TezGoster?key=j_Fjwp4JS4mk97Puqti8rkiC2ELk2iQRp4Md6hu2HSMgdGSsqnEHfw2Ulqyn3nfW